CLINICAL TRIAL: NCT06168448
Title: Non Interventional Study Evaluating the Contribution of a Video to Patient Information Before a Complementary Examination in Infectious Diseases
Brief Title: Contribution of a Video Support to Inform the Patient Before a Complementary Examination in Infectious Diseases
Acronym: AVIEMI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 230351; 2023-A00266-39 (Other: ID-RCB)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Infectious Disease
Keywords: Patient information tool; Understanding of delivered information; Complementary examinations; Video information
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1 : Patients with oral and written information: Group made up of patients hospitalized at that time in the infectious diseases department who met the eligibility criteria set out in the protocol.
  This group of patients will receive the legal oral and written information concerning the additional examination prescribed, as usually delivered by their doctor.
  Interventions: Other: Oral and written information
- Group 2 : Patients with oral and written information + video information: Group made up of patients hospitalized at that time in the infectious diseases department who met the eligibility criteria set out in the protocol.
  This group of patients will receive the legal oral and written information concerning the additional examination prescribed, as usually delivered by their physician, and in addition the video tool will be applied to them.
  Interventions: Other: Oral and written information; Other: Video information
- Group 3 : Caregivers: Nurses and physicians working in the infectious and tropical diseases department.
  This group of caregivers will assess the impact of the intervention on their practice.

INTERVENTIONS:
Other: Oral and written information — Legal oral and written information given by physicians concerning additional examinations
  Groups: Group 1 : Patients with oral and written information; Group 2 : Patients with oral and written information + video information
Other: Video information — Explanatory video applied after physician's formal information
  Groups: Group 2 : Patients with oral and written information + video information

SUMMARY:
The purpose of this study is that a video tool coupled with standardized information can increase the patient's understanding of the information and thus optimize their medical care

DETAILED DESCRIPTION:
Patients admitted to the Infectious and Tropical Diseases Department (MIT) undergo a large number of complementary examinations. In view of their specificity, justified by the often lengthy diagnostic process, as well as by the complexity and diversity of the pathologies, the site of infection and the patient's background (adolescents and adults, migrant patients, immunocompromised patients, Human Immunodeficiency Virus, primary immunodeficiencies, organ transplants, patients with haemopathies, marrow transplants, among others). As a matter of practice, the doctor informs the patient of the prescribed examinations, explaining their purpose and procedure, and outlining any benefits and risks.

The intention is to introduce a tool that complements the information usually provided, and that can be of high quality to improve the patient's perception of understanding. To this end, investigators hypothesize that a tool in video format, built in collaboration with the experience of various technical platforms, could make the experience of understanding information more complete and more accessible to all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* French speaking language
* Hospitalized in the Department of Infectious and Tropical Diseases at Hôpital Necker- Enfants malades
* Prescription, for the first time in its medical history, of one of the following complementary examinations:

  * Bronchial FibroscopyIRM
  * PICC line insertion
  * PET Scanner
* No expressed oral opposition

Exclusion Criteria:

* Patients with dementia or cognitive impairment
* Non-French-speaking patient

Caregivers' inclusion Criteria:

* Caregiver belonging at nurse or doctor's category
* Caregiver working in the Infectious and Tropical Diseases Department at Necker Hospital
* No expressed oral opposition
* Caregivers who are not in contact with patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in the Department of Infectious and Tropical Diseases at Hôpital Necker- Enfants maladies.
  Caregivers working in the Infectious and Tropical Diseases Department at Necker Hospital
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Score of perceived understanding of information before additional examination | up to 7 days
  Measure the patient's perception of comprehension prior to the examination, using a self-assessment Numerical Scale (NRS) defined from zero (no comprehension) to ten (perfect comprehension). The assessment will be collected by a caregiver who is not in charge of the patient, within a maximum of 24 hours after the carried out examination.

SECONDARY OUTCOMES:
Score of perceived understanding of information after additional examination | up to 7 days
  Measure the patient's perception of comprehension after the examination, using a self-assessment Numerical Scale (NRS) defined from zero (no comprehension) to ten (perfect comprehension).
Failure rate of examinations | up to 7 days
  A failure is defined as an examination not performed and/or an examination that cannot be interpreted. The failure is recorded upon return from the examination via the report provided by the technical platform and certified by the physician
Missing elements | up to 7 days
  Collection of elements identified as missing by the patient during the examination. A questionnaire will completed by the patient at his return, in a maximum of 24 hours
Impact on caregivers' knowledge | 1 day
  using a self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LANTERNIER, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Elisabete GOMES-PIRES, Nurse, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants malades, Paris, France